CLINICAL TRIAL: NCT00752622
Title: Optimization of Treatment With Infliximab in a Medical Setting
Brief Title: Treatment With Infliximab in a Medical Setting (Study P05587)
Acronym: OPTIMIST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Factors that led to termination: recruitment challenges and a lower incidence of flares than estimated, causing a high risk of the study being underpowered.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05587
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shortened interval (Experimental): Infliximab 5 mg/kg, then Infliximab 5 mg/kg every 6 weeks
  Interventions: Biological: Infliximab 5 mg/kg; Biological: Infliximab 5 mg/kg every 6 weeks
- Increased dose (Experimental): Infliximab 5 mg/kg, then Infliximab 7 mg/kg every 8 weeks
  Interventions: Biological: Infliximab 5 mg/kg; Biological: Infliximab 7 mg/kg every 8 weeks

INTERVENTIONS:
Biological: Infliximab 5 mg/kg — Participants received Infliximab 5 mg/kg intravenously (IV) at weeks 0, 2 and 6 during the induction phase. At Week 10, those who were in clinical response received further treatment every 8 weeks during the observational phase
  Other Names: Remicade; SCH 215596
Biological: Infliximab 5 mg/kg every 6 weeks — Participants with loss of response in the observational phase were randomized at entry into the interventional phase received 5 mg/kg IV every 6 weeks (shortened interval group)
  Arms: Shortened interval
Biological: Infliximab 7 mg/kg every 8 weeks — Participants with loss of response in the observational phase were randomized at entry into the interventional phase received 7 mg/kg IV every 8 weeks (increased dose group)
  Arms: Increased dose

SUMMARY:
This is an open-label, interventional study where a subset of participants will be randomized to one of two treatment-optimization strategies. Participants with moderate to severe Crohn's disease (CD) will receive induction treatment comprised of 3 infusions of infliximab at Weeks 0, 2, and 6. The participants will be evaluated at Week 10. Participants who are in clinical response will enter the observational phase of the study where they will receive standard of care treatment, as per the infliximab product monograph. Participants who lose response, may qualify for entry into the interventional phase of the study, where they will be randomized to one of the following treatment-optimization arms: 1) dose increase: infliximab 7 mg/kg, every 8 weeks or 2) shortened interval: infliximab 5 mg/kg every 6 weeks.

Note: Due to early study termination, no statistical analysis was performed for the interventional part of this study, therefore, endpoints dedicated to this phase of the study have not been analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >=18 years of age
* Moderate to severe CD (Crohn's Disease Activity Index [CDAI] >= 220 and <= 450)
* CD of at least 3 months duration confirmed within the past 2 years by radiography and/or endoscopy
* Biologic-naïve
* If using 5-Aminosalicylic Acid (5-ASA), there must be at least 4 weeks of stable dosage prior to screening
* If using azathioprine or 6-mercaptopurine, the start date must be at least 3 months prior to screening and the dose must be stable for at least 6 weeks prior to screening
* If using methotrexate, the participant must have been using methotrexate with a stable dosage of at least 6 weeks prior to screening
* Participants must be off corticosteroids or on a stable dose of corticosteroids for at least 2 weeks prior to enrollment. The maximal daily dose of corticosteroids at baseline must not exceed 30 mg of prednisone equivalent
* Participants are considered eligible according to the following tuberculosis (TB) screening criteria:

  * Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination
  * Have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study medication
  * Within 3 months prior to the first administration of study medication, either have negative OR have a newly identified positive diagnostic TB test result (defined as at least 1 positive tuberculin skin test) during screening in which active TB has been ruled out, and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study medication
  * Participants must have had a chest X-ray within 3 months prior to screening with no evidence of current or old active TB
* Participants' screening and baseline clinical laboratory tests (complete blood count [CBC], blood chemistries, and urinalysis) must be within the following parameters:

  * Hemoglobin >=10 g/dL (100 g/L)
  * White blood cells (WBCs) >=3.5 x 109/L
  * Neutrophils >=1.5 x 10^9/L
  * Platelets >=100 x 10^9/L
  * Serum creatinine <1.5 mg/dL (or <133 μmol/L)
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, and gammaglutamyltransferase <=1.5 x upper limit of normal (ULN);
  * Total bilirubin <=1 x ULN
* Antibiotics for the treatment of CD (e.g., ciprofloxacin and metronidazole) must have been discontinued at least 3 weeks prior to screening
* Participants must be free of any clinically significant condition or situation, other than CD that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study
* Participants are willing and able to adhere to the study visit schedule and other protocol requirements
* Participants are capable of providing written informed consent, which must be obtained prior to conducting any protocol-specified procedures
* Sexually-active women of child-bearing potential must agree to use a medically accepted method of contraception prior to screening, while receiving protocol specified medication, and for 6 months after stopping the medication
* Women of child-bearing potential who are not currently sexually active must agree to use a medically accepted method of contraception should they become sexually active while participating in the study
* Female participants of childbearing potential must have a negative serum pregnancy test (beta-hCG) at screening
* have an increased Harvey-Bradshaw Index (HBI) score >=3 points over the week 10 evaluation score and a CDAI score >=175
* have received regular infusions of Infliximab (IFX) every 8 weeks during the observational phase with a maximum interval of no more than 10 weeks between each infusions
* having previous doses of IFX of >= 4.7 mg/kg

Exclusion Criteria:

* Are pregnant or plan to become pregnant during the study period; participants who are breast feeding
* Have been treated with excluded drugs prior to entry: any biological or anti- Tumor necrosis factor (anti-TNF) agent such as infliximab, adalimumab, certolizumab, etanercept, pentoxifylline, or thalidomide
* Have had a serious infectious disease in the 8 weeks prior to entry
* Have active perianal fistulas and a Perianal disease activity index (PDAI) score >10
* Have presumed fibro-stenotic stricture or acute bowel obstruction
* Have had live vaccination in the 6 weeks prior to entry
* Have known intolerance to study drug
* Have a history of myocardial infarction, congestive heart failure, coronary artery disease, or arrhythmias in the last 6 months
* Have a history of malignancy (within the past 5 years) with the exception of carcinoma in situ of the cervix or localized basal cell skin cancer that have been adequately treated
* Have a history of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease
* Have a history of demyelinating disease such as multiple sclerosis
* Have a positive test for human immunodeficiency virus (HIV), hepatitis B virus (HBV) surface antigen, or hepatitis C virus (HCV) antibody
* Have renal, hepatic, hematological, cardiovascular, pulmonary, neurological, psychiatric, immunologic, gastrointestinal, endocrine, or other diseases if they are clinically significant. (A clinically significant disease is defined as one which in the opinion of the investigator can put the participants at risk because of participation in the study or a disease which can influence the participant's ability to participate in the study or affect the results of the

study)

* Have clinically significant abnormal laboratory test results, unless regarded by the investigator as related to CD
* Have a history of alcohol or drug abuse
* Are unable to comply with the protocol
* Have any clinically significant findings in the physical examination that, in the investigator's judgment, may interfere with the study evaluation or affect participant safety
* Are in a situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study
* Are participating in any other clinical study(ies) except for registries
* Are on the staff, affiliated with, or a family member of the staff personnel directly involved with this study
* Are allergic to or have sensitivity to the study drug or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 100 enrolled participants, 2 participants experienced a protocol violation that excluded them from the Eligible (ELIG) population, thus, the ELIG population comprised of 98 participants.
  Due to early study termination, all 8 randomized participants received at least one infusion of interventional treatment, but none completed the trial.
Groups:
- Infliximab: Infliximab 5mg/kg intravenously (IV) at weeks 0, 2 and 6 during the induction phase and every 8 weeks during the observational phase and either 5mg/kg every 6 weeks or 7mg/kg every 8 weeks as determined by randomization at entry into the interventional phase.
Period: Induction Phase
Arm/Group | Infliximab
Started | 100 (The ELIG population comprised of 98 participants)
Completed | 65
Not Completed | 35
Not completed — Adverse Event | 3
Not completed — Other | 3
Not completed — Non-responder | 14
Not completed — Withdrawal by Subject | 1
Not completed — Premature study termination | 14
Period: Observational Phase
Arm/Group | Infliximab
Started | 65
Completed | 22 (14 completed without loss of response 8 had loss of response & randomized into interventional phase)
Not Completed | 43
Not completed — Premature Study Termination | 36
Not completed — Non-responder | 2
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Other | 2
Period: Interventional Phase
Arm/Group | Infliximab
Started | 8 (5 participants randomized into increased dose group and 3 randomized into shortened interval group)
Completed | 0 (8 participants received at least 1 infusion of interventional treatment, but none completed trial)
Not Completed | 8
Not completed — Non-responder | 2
Not completed — Physician Decision | 1
Not completed — Premature Study Termination | 5

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — The mean age at baseline within the population of all eligible (ELIG) participants (Overall= 98).
  years | 38.4 (13.16)
Sex/Gender, Customized [Number; unit: participants]
  Female | 54
  Male | 44
  Excluded from analysis | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Clinical Response Using the Crohn's Disease Activity Index (CDAI) at Week 24 in the Interventional Phase
Description: The CDAI incorporates 8 items that are indicators of disease severity. Scores range from 0 to ~600; higher scores indicate worse disease activity. Participants with scores below 150 have inactive disease whereas those with scores above 450 are considered critically ill. Participants provided completed CDAI diary cards and were considered as responders in the interventional phase if their CDAI score at week 24 was decreased by 70 points or greater over their CDAI score at randomization into the interventional phase, or if their week 24 CDAI score is <= 150. Baseline is value at randomization.
Time Frame: Baseline and Week 24 of the Interventional phase
Population: Due to the early termination of the study, no participants completed the Interventional phase.
Arm/Group | Infliximab
Number analyzed (Participants) | 0

2. Primary Outcome: Mean Change From Baseline in Harvey-Bradshaw Index (HBI)
Description: Mean change in HBI score from Baseline to Week 10, 30, and 54. HBI score consists of clinical parameters: general well-being (0-4), abdominal pain (0-3), number of liquid stools per day, abdominal mass (0-3), and complications (score 1 per item). Total score is the sum of individual parameters. Minimum score is 0 and no pre-specified maximum score as it depends on the number of liquid stools. Lower scores indicate better well being. Clinical response/ long-term response is defined as a decrease by 3 or more points from baseline value. Loss of response is defined as an increase of >= 3 points.
Time Frame: Baseline and Evaluation Week 10, Week 30 and Week 54 of the Observational Phase
Population: The eligible (ELIG) population comprised a subset of the enrolled (ENR) population who were not associated with an important protocol violation and who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 98
score on a scale
  Baseline (n= 98) | 9.5 (3.23)
  Change at Week 10 (n= 81) | -5.88 (3.890)
  Change at Week 30 (n= 37) | -7.19 (2.998)
  Change at Week 54 (n= 15) | -7.93 (3.173)
Statistical Analysis 1: Comparison: Infliximab; Comparison of Infliximab from Induction baseline to evaluation Week 10; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Infliximab; Comparison of Infliximab from Induction baseline to Week 30 of the Observational Phase; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Infliximab; Comparison of Infliximab from Induction baseline to Week 54 of the Observational Phase; Test type: Superiority or Other; p < .0001, t-test, 2 sided

3. Secondary Outcome: Number of Participants That Required Treatment Optimization in the Observational Phase
Description: Participants required treatment-optimization if:
  * Disease progression/lack of response after entering observational phase; or
  * Participant was successfully randomized into the interventional phase
  The definition of loss of response was as follows:
  - An increased HBI score >= 3 points over the week 10 evaluation score and a CDAI score >= 175.
  Despite:
  * having received regular infusions of infliximab every 8 weeks during the observational phase with a maximum interval of no > 10 weeks between each infusion, and
  * having received previous doses of infliximab of >= 4.7 mg/kg.
Time Frame: Week 54 in the Observational Phase
Population: The eligible (ELIG) population comprised a subset of the enrolled (ENR) population who were not associated with an important protocol violation and who received at least one dose of study medication. Of the 98 participants in the ELIG population, 65 participants entered the observational phase.
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 65
Participants | 10

4. Secondary Outcome: Number of Participants Who Had a Clinical Response Using the CDAI at Weeks 14-16 and 48 in the Interventional Phase
Description: The CDAI incorporates 8 items that are indicators of disease severity. Scores range from 0 to ~600; higher scores indicate worse disease activity. Participants with scores below 150 have inactive disease whereas those with scores above 450 are considered critically ill.
  Clinical response was defined as a 70-point reduction in CDAI score from randomization into the interventional phase or CDAI < 150 at week 14-16 and 48 in the Interventional Phase. Baseline is value at randomization.
Time Frame: Baseline and Weeks 14-16 and 48 in the Interventional Phase
Population: Due to the early termination of the study, no participants completed the Interventional phase.
Arm/Group | Infliximab
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Had a Clinical Response Using the CDAI-100 at Weeks 14-16, 24 and 48 in the Interventional Phase
Description: The CDAI incorporates 8 items that are indicators of disease severity. Scores range from 0 to ~600; higher scores indicate worse disease activity. Participants with scores below 150 have inactive disease whereas those with scores above 450 are considered critically ill.
  Clinical response was defined as a 100-point reduction in CDAI score from randomization into the interventional phase or CDAI < 150 at weeks 14-16, 24 and 48 in the Interventional Phase. Baseline is value at randomization.
Time Frame: Baseline and Weeks 14-16, 24 and 48 in the Interventional Phase
Population: Due to the early termination of the study, no participants completed the Interventional phase.
Arm/Group | Infliximab
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants Who Had Clinical Remission in the Interventional Phase
Description: The CDAI incorporates 8 items that are indicators of disease severity. Scores range from 0 to ~600; higher scores indicate worse disease activity. Participants with scores below 150 have inactive disease whereas those with scores above 450 are considered critically ill.
  Clinical remission was defined as CDAI < 150 at weeks 14-16, 24 and 48 in the Interventional Phase.
Time Frame: Weeks 14-16, 24 and 48 in the Interventional Phase
Population: Due to the early termination of the study, no participants completed the Interventional phase.
Arm/Group | Infliximab
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Who Had Clinical Remission Off Steroids in the Interventional Phase
Description: Number of participants who were in clinical remission and off systemic corticosteroids at visit.
  The CDAI incorporates 8 items that are indicators of disease severity. Scores range from 0 to ~600; higher scores indicate worse disease activity. Participants with scores below 150 have inactive disease whereas those with scores above 450 are considered critically ill. Clinical remission was defined as CDAI < 150 at weeks 14-16, 24 and 48 in the Interventional Phase.
Time Frame: Weeks 14-16, 24 and 48 in the Interventional Phase
Population: Due to the early termination of the study, no participants completed the Interventional phase.
Arm/Group | Infliximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Enrolled Analysis population (ENR). The ENR population comprised all participants enrolled into the Induction Phase of the protocol and were included in the safety population.
Groups:
- Infliximab 5 mg/kg Then Not Randomized: Infliximab 5 mg/kg IV at weeks 0, 2 and 6 during the induction phase as well as every 8 weeks during the observational phase. Participants who were further randomized into the interventional phase are not included in this reporting group; therefore, of the 100 enrolled participants, 92 participants were included in this safety reporting group.
- Infliximab 5 mg/kg Then Randomized: Infliximab 5 mg/kg IV at weeks 0, 2 and 6 during the induction phase as well as every 8 weeks during the observational phase. Participants were then randomized to receive 5 mg/kg every 6 weeks (shortened interval group) or 7 mg/kg every 8 weeks (increased dose group) at entry into the interventional phase. This reporting group included 3 participants randomized into the shortened interval group and 5 participants randomized into the increased dose group.
Arm/Group | Infliximab 5 mg/kg Then Not Randomized | Infliximab 5 mg/kg Then Randomized
Serious Adverse Events (participants affected / at risk) | 7/92 | 3/8
Other Adverse Events (participants affected / at risk) | 42/92 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg Then Not Randomized (N=92) | Infliximab 5 mg/kg Then Randomized (N=8)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's Disease (Gastrointestinal disorders) | 2 (2) | 1 (2)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infusion Related Reaction (General disorders) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pelvic Abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg Then Not Randomized (N=92) | Infliximab 5 mg/kg Then Randomized (N=8)
Abdominal Pain (Gastrointestinal disorders) | 7 (11) | 1 (1)
Abdominal Tenderness (Gastrointestinal disorders) | 4 (4) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Crohn's Disease (Gastrointestinal disorders) | 5 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (11) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (7) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (11) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 2 (2)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 10 (14) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early study termination, no statistical analysis was performed for the interventional part of this study, therefore, endpoints dedicated to this phase of the study have not been analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication of results obtained in this study, written permission is required. Draft manuscripts, abstracts & presentations should be submitted for review & approval. Schering-Plough Canada will retain the ownership of the data obtained in this study. Authorship of publications resulting from this study should accurately reflect the academic contribution of individuals to the design and implementation of the study, analysis of the data and preparation of the manuscript.